CLINICAL TRIAL: NCT02822469
Title: Thermograph Evaluation of Masticatory Muscles Pre and Post Indirect Physiotherapeutic Treatment in TMD Subjects: A Randomized, Placebo-controlled Study
Brief Title: Thermograph Evaluation of Masticatory and Cervical Muscles After Physiotherapeutic Treatment in Tmd Subjects
Acronym: TEMCMAPTTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daniela Ap. Biasotto-Gonzalez (Other)
Responsible Party: Sponsor-Investigator, Daniela Ap. Biasotto-Gonzalez, DR, University of Nove de Julho
Organization: University of Nove de Julho (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2YEH1984
Record Dates: First submitted 2016-06-23; First posted 2016-07-04 (Estimated); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Temporomandibular Joint Dysfunction
Keywords: TMD Infrared Thermography Physical Therapy Modalities
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manual Therapy Treatment Group (Experimental): Severe and Moderate TMD patients who filled the inclusion criteria who will receive the Manual Therapy Treatment
  Interventions: Other: Manual Therapy Treatment
- Placebo Ultrasound Treatment Group (Placebo Comparator): Severe and Moderate TMD patients who filled the inclusion criteria who will receive the Placebo Treatment.
  Interventions: Device: Placebo Ultrasound

INTERVENTIONS:
Other: Manual Therapy Treatment — Treatment starts with 10 deep breathing movements for global relaxation. The anterior and posterior neck muscles, shoulder girdle and subdiaphragmatic will be addressed with myofascial techniques repeated 10 times in each stroke. The cervical spine will be pulled in the longitudinal direction. The draw will be held 1 time, lasting 1 minute. The thoracic region will receive mobilization technique in the anteroposterior direction,10 repeated movements involving all thoracic segment.
  The treatment will be applied previously trained therapists, 4 weeks, 2 times a week, totaling eight sessions. The treatment time per session is about 25 minutes.
  Arms: Manual Therapy Treatment Group
Device: Placebo Ultrasound — A detuned pulsed ultrasound will be applied to regions of the muscles around the shoulder girdle and anterior posterior cervical, for 25 minutes (2.5 minutes in each zone ). The device will be used with the internal cables disconnected for the placebo effect . However, you can handle it and adjust the doses and alarms as it is connected in order to simulate clinical practice and increase the credibility of the use of this device in the voluntary . The placebo treatment will be applied by previously trained therapists. Treatment will have 4 weeks, 2 times a week, totaling eight sessions.
  Arms: Placebo Ultrasound Treatment Group

SUMMARY:
Background: Different therapeutic approaches have been proposed for the treatment of TMD. Myofascial and joint techniques, exercises, intraoral devices, thermal, electro and phototherapy applications, are among the most common. The combination of local treatments and adjacent structures such as the cervical region have also been studied in this area. It is believed that the anatomic proximity, neuronal interconnections and convergent afferents from the trigeminal and cervical areas can lead the understanding of the relationship of these structures. In order to assess the effects of these different forms of treatment studies have used different resources such as diagnostic imaging and biological signals, in order to complement the clinical diagnosis. Infrared thermography has been one of the resource assessment in the literature and it is interesting and stands out from other methods because it is functional, non-invasive and inexpensive.

Purpose: To evaluate the thermograms concerning the masseter and anterior temporal muscles, severity, pain, range of mandibular motion and neck disability in TMD patients, before and after physical therapy applied to the cervical and thoracic regions.

Methods: This is a randomized, placebo-controlled study, designed to evaluate the effects of indirect treatment on the thermography of the masticatory muscles, severity, pain, range of motion and neck disability in individuals with TMD. These will be randomized and allocated into two groups: GA (intervention) and GB (placebo) and assessed as: Diagnostic Criteria for Temporomandibular Research Disorders (RDC/TMD), Fonseca´s Anamnesic Index (FAI), Thermography, EVA, IDD-CF, Pachymetry and Neck Disability Index (NDI).

Statistical analysis: The temperature of the orofacial region, acquired through thermography is considered the primary endpoint and as a secondary endpoint will be the evaluation of the severity according to FAI, pain by VAS and IDD-CF, the range of mandibular motion by pachymetry and neck disability by NDI.

Statistical analysis: The normality of the data will be verified using the Kolmogorov-Smirnov test, which will be expressed as mean and standard deviation and/or median and interquartile range. Repeated measures analysis of variance of two factors, post hoc Bonferroni will be used for inter and intra-group comparisons. The significance level of p≤0.05 is set.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, study designed to evaluate the thermograms concerning the masseter and anterior temporal muscles, severity, pain, range of mandibular motion and neck disability in TMD patients, before and after physical therapy applied to the cervical and thoracic regions.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45 years;
* presence of pain in the facial region in the last 6 months;
* diagnosis of myofascial pain (I) and/or disc displacement (IIa and IIb) determined by the DRC/TMD; Moderate DTM Record carrier or determined by Fonseca Anamnesic Index.

Exclusion Criteria:

* A history of trauma/cervical surgery and/or craniofacial;
* Neurological disorders;
* cervical disc disease;
* degenerative diseases of the spine;
* systemic diseases;
* diagnosis of fibromyalgia;
* prior treatments for TMD for the last 3 months;
* orthodontic treatment/orthopedic in progress;
* continuous use of analgesics, anti-inflammatories, anxiolytics and/or antidepressants;
* BMI> 25 kg / m2;
* pregnancy.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Changes in Skin Temperature | Baseline and 4 weeks
  Measured by the Infrared thermographic digital camera

SECONDARY OUTCOMES:
Changes in TMD severity | Baseline and 4 weeks
  Measured by Fonseca´s Anamnesic Index
Changes in Neck disability | Baseline and 4 weeks
  Measured by the Neck Disability Index
Changes in Pain incapacity | Baseline and 4 weeks
  Measured by the IDD-CF
Changes in Movement Range of Motion (Opening) | Baseline and 4 weeks
  Measured using a pachymeter (mean values of 3 opening measures)
Changes in Referred Pain | Baseline and 4 weeks
  Measured by Visual Analogic Scale

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Ap Biasotto-Gonzalez, PHD, Study Chair — Study Principal Investigator - Universidade Nove de Julho
Locations (1):
- University of Nove de Julho, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No